CLINICAL TRIAL: NCT05789485
Title: Dose-response of Aerobic Training During Chemotherapy for Gastrointestinal Cancers
Brief Title: A Study on the Effects of Exercise on Side Effects From Treatment for Gastrointestinal Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-164
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Cancer
Keywords: Exercise; 22-164
MeSH Terms: conditions — Gastrointestinal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients and investigators will be blinded to results during study conduct.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 90 min/wk (Experimental): AT will consist of individualized walking delivered up to 7 times per week to achieve a cumulative total duration of: Arm 1: 90 min/wk. AT therapy within each arm will follow a non-linear (i.e., AT dose is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule delivered during chemotherapy. Supervised AT will be monitored using TeleEx.
  Interventions: Behavioral: structured treadmill walking
- 150 mins/wk (Experimental): AT will consist of individualized walking delivered up to 7 times per week to achieve a cumulative total duration of: Arm 2: 150 min/wk. AT therapy within each arm will follow a non-linear (i.e., AT dose is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule delivered during chemotherapy. Supervised AT will be monitored using TeleEx.
  Interventions: Behavioral: structured treadmill walking
- 300 mins/wk (Experimental): AT will consist of individualized walking delivered up to 7 times per week to achieve a cumulative total duration of: Arm 3: 300 min/wk. AT therapy within each arm will follow a non-linear (i.e., AT dose is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule delivered during chemotherapy. Supervised AT will be monitored using TeleEx.
  Interventions: Behavioral: structured treadmill walking

INTERVENTIONS:
Behavioral: structured treadmill walking — Three doses of AT (i.e., 90, 150, or 300 mins/week) will be tested. All doses will consist of individualized walking delivered up to 7 times per week delivered throughout treatment.

SUMMARY:
The purpose of this study is to find the level of aerobic exercise (AT) that is practical, is safe, and has positive effects on the body that may reduce the side effects of therapy. The study will also look at the way the body responds to exercise and whether there are differences in treatment. This will include looking at the highest treatment dose participants receive, how many people stop, delay, or reduce the treatment, and whether additional medication is needed to treat side effects of therapy.

DETAILED DESCRIPTION:
Study staff will also confirm remote training feasibility including items such as access to Wi-Fi and a treadmill for the study duration. During the feasibility assessment, if the participant is determined to not have access to Wi-Fi, we will offer a tablet with cellular capabilities. If patients do not have access to a treadmill, ExOnc staff may coordinate access to a fitness facility local to the participant, to facilitate treadmill access for the study duration. Fitness facility access will be provided through Wellhub, a service that allows use of nearby gyms and studios through a single app- based solution.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Diagnosed with colorectal or esophago/gastric solid tumors as defined by one of the following:

  * Histological confirmation
  * As per standard of care imaging
* Scheduled to receive neoadjuvant chemotherapy or chemotherapy for newly diagnosed metastatic disease
* Performing ≤90 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures
* Cleared for exercise participation as per screening clearance via the Physical Activity Readiness Questionnaire

Exclusion Criteria:

* Enrollment onto any other lifestyle interventional investigational study, except interventions determined by the PI not to confound study outcomes
* Receiving treatment for any other diagnosis of invasive cancer
* Mental impairment leading to inability to cooperate
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
proportion of patients achieving (ratio of delivered to planned treatment) RDI ≥ 90% | 5 years
  RDI (%) will be calculated as the ratio of delivered to planned dose intensity (delivered dose intensity/planned dose intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Hartford Healthcare Alliance (Data Collection Only), Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm